CLINICAL TRIAL: NCT05135104
Title: Non-Interventional, National Study Of Real-World Evidence In Estrogen Receptor Positive, Her2 Negative Metastatic Breast Cancer Patients Treated With Palbociclib During a 2.5 Years Follow-Up Period
Brief Title: Study Of Real-World Evidence In Patients Treated With Palbociclib During a 2.5 Years Follow-Up Period
Acronym: PALBO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asociatia Oncohelp - Centrul de Oncologie Oncohelp (Other)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Other Study IDs: PALBO01/2021
Record Dates: First submitted 2021-11-01; First posted 2021-11-26 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; Metastatic Breast Cancer; Her2 Negative Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Palbociclib — Palbociclib, an orally active pyridopyrimidine, is a potent and highly selective reversible inhibitor of CDK 4 and CDK6. The compound prevents cellular DNA synthesis by prohibiting progression of the cell cycle from G1 into the S phase. Specifically, Palbociclib inhibits CDK4/6-catalyzed phosphorylation of the retinoblastoma protein (Rb), which is required for cell division.
  Palbociclib has selectivity for CDK4/6, with little or no activity against a large panel of 274 other protein kinases including other CDKs and a wide variety of tyrosine and serine/threonine kinases.
  Therapeutic indications:
  Palbociclib is indicated for the treatment of hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative locally advanced or MBC:
  * in combination with an aromatase inhibitor;
  * in combination with fulvestrant in women who have received prior endocrine therapy.
  Other Names: Ibrance

SUMMARY:
PALBO is a Non-Interventional, National Study Of Real-World Evidence In Estrogen Receptor Positive, Her2 Negative Metastatic Breast Cancer Patients Treated With Palbociclib During A 2.5 Years Follow-Up Period. The primary objective is to identify pathological and clinical features of MBC that is associated with Palbociclib's best efficacy, measured by response rate (overall response rate, duration of response and best clinical response), progression free survival and OS. Safety of Palbociclib will also be evaluated.

DETAILED DESCRIPTION:
Metastatic breast cancer (MBC) is the most advanced stage of breast cancer, where the disease has spread to distant sites beyond the axillary lymph nodes. At European level, MBC occurs in up to 20-30 percent of women diagnosed with early-stage breast cancer. At regional level, there are variations in newly diagnosed patients who present with metastatic disease. In high income countries fewer than 8% of patients are initially diagnosed with MBC, while the highest burden of MBC is carried by low and middle-income countries where up to 60% are initially diagnosed with MBC. Currently, the median overall survival for patients with MBC is approximately 2 to 3 years in developed countries, but lower in developing countries. In Romania, 8900 new cases of BC are diagnosed every year, with 80% being diagnosed in an advance stage of the disease (II, III, IV). Furthermore, after initial BC treatment, approximately 50% will develop MBC.

Cyclin-dependent kinase (CDK) 4/6 inhibitors (Palbociclib, ribociclib and abemaciclib) are now standard of care for the treatment of advanced hormone receptor positive (HR+) and HER2 negative (HER2-) breast cancer.

On 09 November 2016, the EC has approved IBRANCE® (Palbociclib) as the first CDK 4/6 inhibitor, to be used in combination with letrozol as first-line or in combination with fulvestrant in women who have received prior endocrine therapy, based on the results of PALOMA-1, PALOMA-2 and PALOMA-3 study results. Other phase III randomized trials have been reported and confirmed the efficacy of CDK4/6 inhibition in both first-line and endocrine resistant settings.

Palbociclib®, an orally active pyridopyrimidine, is a potent and highly selective reversible inhibitor of CDK 4 and CDK6. The compound prevents cellular DNA synthesis by prohibiting progression of the cell cycle from G1 into the S phase. Specifically, Palbociclib inhibits CDK4/6-catalyzed phosphorylation of the retinoblastoma protein (Rb), which is required for cell division.

Palbociclib® has selectivity for CDK4/6, with little or no activity against a large panel of 274 other protein kinases including other CDKs and a wide variety of tyrosine and serine/threonine kinases.

An approximate number of 650 patients will be included in the present study which will take place on national level in 6 sites in Romania.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women and men (≥ 18 years of age) with proven initial diagnosis of breast cancer with evidence of loco-regional recurrent or metastatic disease not amenable to resection or radiation therapy.
2. Documentation of histologically or cytologically confirmed diagnosis of breast cancer with IHC of estrogen receptor (ER) expression > 1% and/or progesterone receptor (PR) expression >1 % breast cancer based on local laboratory results.
3. Scoring of 0 or 1+ for HER2 protein expression by a validated immunohistochemistry assay or +1/+2 with negative HER2 amplification FISH/ISH ratio lower than 1.8 or HER2 gene copy less than 4.0.
4. Eligible subjects must have undergone a treatment with Palbociclib for at least 3 months.
5. Measurable or evaluable disease as defined per modified Response Evaluation Criteria in Solid Tumours (mRECIST) V1.1 criterion (at least 2 entries).
6. Premenopausal or postmenopausal status.

6.1 Patients who are not postmenopausal must have undergone a treatment with LHRH agonist.

6.2 Postmenopausal status is defined as:

1. prior bilateral surgical oophorectomy, or
2. spontaneous cessation of regular menses for at least 12 consecutive months
3. in case of doubt serum estradiol <20 umol/l and follicle stimulating hormone (FSH) levels >15 IU/L.

Exclusion Criteria:

1. Subjects with advanced, symptomatic, visceral spread, such as patients with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50% liver involvement).
2. Palbociclib treatment as part of a clinical trial or prescription prior to market approval (Nov 2016).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects aged 18 years and older with a confirmed diagnosis of Estrogen Receptor Positive, HER2 Negative MBC. Eligible subjects must have undergone a treatment with Palbociclib for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) in subjects participating in the clinical investigation [ Time Frame: 2.5 years] | 2.5 years
  DCR will be calculated per modified Response Evaluation Criteria in Solid Tumours (mRECIST) V1.1 criterion, as the proportion of patients with best overall response to protocol therapy of complete response (CR), partial response (PR) or stable disease (SD) that is maintained for at least 12 weeks.
Overall Survival (OS) investigation [ Time Frame: 2.5 years] | 2.5 years
  OS will be defined as the elapsed time from the enrolment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will at 1, 2 and 3 months until death or withdrawal of consent from the study.
Objective Response Rate (ORR) investigation [ Time Frame: 2.5 years] | 2.5 years
  ORR will be defined as the proportion of the patients with a confirmed CR or PR, as per mRECIST V1.1 criterion.
Duration of Response (DOR) investigation [ Time Frame: 2.5 years] | 2.5 years
  DOR will be defined as the elapsed time from documented tumour response to documented disease progression.

SECONDARY OUTCOMES:
The medium duration of the treatment with Palbociclib in combination with aromatase inhibitors (AI) in first-line and with fulvestrant in second-line | 2.5 years
  The first secondary objective of our study is to identify the medium duration of the treatment with aromatase inhibitors (AI) in first-line and with fulvestrant in second-line.
The Clinical Benefit Rate (CBR), defined as the proportion of patients with no disease progression after 6 months of therapy. | 6 months after therapy start
  The second secondary objective of our study is to identify the Clinical Benefit Rate (CBR), defined as the proportion of patients with no disease progression after 6 months of therapy.
PFS in a selected subgroup with KI67 mutation | 2.5 years
  Exploratory variable
PFS in a selected subgroup of subjects with lower levels of HER2 expression (HER2-low) defined as HER2 immunohistochemistry 1+ or 2+, but FISH negative | 2.5 years
  Exploratory variable
PFS in lobular/ductal/other histological subtypes | 2.5 years
  Exploratory variable
PFS in a selected subgroup with Luminal B subtype | 2.5 years
  Exploratory variable

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Marinela Oprean, MD, Principal Investigator — ASOCIATIA ONCOHELP - CENTRUL DE ONCOLOGIE ONCOHELP, DEPARTMENT OF MEDICAL ONCOLOGY
Locations (7):
- Romania (7):
  - Asociatia Oncohelp - Centrul de Oncologie Oncohelp, Timișoara, Timiș County
  - Spitalul Clinic de Obstetrică Și Ginecologie Filantropia, Bucharest
  - Institutul Oncologic "Prof. Dr I. Chiricuta", Cluj-Napoca
  - Spitalul Clinic Județean de Urgență Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie "Sf. Nectarie", Craiova
  - Institutul Regional de Oncologie, Iași
  - Spitalul Clinic Județean de Urgență Oradea, Oradea